CLINICAL TRIAL: NCT00026078
Title: Docetaxel (DTX) - Ifosfamide (IFX) As First Line Chemotherapy In Metastatic Breast Cancer
Brief Title: Docetaxel and Ifosfamide in Treating Women With Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Grupo Oncologico Cooperativo del Sur (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: GOCS-02-BR-01; CDR0000068969 (Registry Identifier: PDQ (Physician Data Query)); NCI-V01-1670
Record Dates: First submitted 2001-11-09; First posted 2003-01-27 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2006-11

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Ifosfamide

INTERVENTIONS:
Drug: docetaxel
Drug: ifosfamide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of docetaxel and ifosfamide in treating women who have metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of docetaxel and ifosfamide as first-line chemotherapy in women with metastatic breast cancer.
* Determine the response rate and duration of response of patients treated with this regimen.
* Determine the time to treatment failure and survival of patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.
* Determine the quality of life of patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive docetaxel IV over 1 hour on day 1 and ifosfamide IV over 1 hour (beginning 1 hour after docetaxel infusion) on days 1-3. Treatment continues every 4 weeks in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, every month during study, and then every 3 months after completion of study.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 15-42 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic breast cancer
* Bidimensionally measurable lesions

  * The following are not considered measurable:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Inflammatory breast disease
    * Lymphangitis cutis/pulmonis
* Disease progression after hormonal therapy allowed provided at least 1 month since last therapeutic manipulation
* No CNS metastases
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 21 to 75

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* ECOG 0-2 OR
* Zubrod 0-2

Life expectancy:

* More than 12 weeks

Hematopoietic:

* WBC at least 4,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 11 g/dL

Hepatic:

* Bilirubin no greater than 1.25 times upper limit of normal (ULN)
* SGOT no greater than 1.25 times ULN

Renal:

* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No history of congestive heart failure
* No myocardial infarction within the past 6 months
* No active ischemic heart disease
* No uncontrolled hypertension

Other:

* Not pregnant
* No other prior or concurrent malignancy except properly treated basal cell skin cancer or carcinoma in situ of the cervix
* No other medical or psychiatric diseases that would preclude study
* No geographical situation that would preclude study
* No history of alcohol abuse

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior adjuvant chemotherapy including ifosfamide or docetaxel
* No prior systemic chemotherapy for metastatic breast cancer

Endocrine therapy:

* See Disease Characteristics
* No concurrent corticoids, gestagens, or androgens unless strictly indicated

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No concurrent drinks containing caffeine or alcohol

Ages: 21 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2001-03

PRIMARY OUTCOMES:
Response rate

SECONDARY OUTCOMES:
Time to treatment failure
Duration of response
Survival
Toxicity as assessed by CTC version 2.0
Quality of life as assessed by Schipper's Functional Living Index - Cancer

CONTACTS AND LOCATIONS:
Overall Officials: Bernardo A. Leone, MD, Study Chair — Unidad Oncologica Del Neuquen
Locations (8):
- Argentina (7):
  - Grupo Oncologico Cooperativo del Sur, Bahía Blanca, Buenos Aires
  - Policlinica Privada Instituto De Medicina Nuclear, Bahía Blanca, Buenos Aires
  - St. Joseph Medical Center, Manuel B. Gonnet, Buenos Aires
  - Sanatorio Santa Rosa S.R.L., Santa Rosa, La Pampa Province
  - Unidad Oncologica Del Neuquen, Neuquén, Neuquén Province
  - C.R I O., Mar del Plata
  - Centro Oncologico Tres Arroyos, Tres Arroyos
- Centro Medico Nacional de Occidente, Guadalajara, Jalisco, Mexico